CLINICAL TRIAL: NCT02305030
Title: Effect of Opicapone at Steady State on Warfarin Pharmacokinetics in Healthy Volunteers
Brief Title: Effect of Opicapone at Steady State on Warfarin Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-127
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIA 9-1067 / Warfarin (Experimental): BIA 9-1067 capsules of 25 mg or 50 mg Warfarin capsules of 5 mg
  Interventions: Drug: BIA 9-1067; Drug: Warfarin

INTERVENTIONS:
Drug: BIA 9-1067
  Other Names: OPC, Opicapone
Drug: Warfarin
  Other Names: Uniwarfin

SUMMARY:
Single-centre, open-label, fixed-sequence design consisting of 2 periods separated by a washout period of at least 14 days.

DETAILED DESCRIPTION:
Single-centre, open-label, fixed-sequence design consisting of 2 periods separated by a washout period of at least 14 days. In Period 1, a single dose of 25 mg warfarin was administered alone. In Period 2, subjects received 475 mg OPC, on Day 1 and D2 followed by 50 mg OPC once daily for 5 days (D3 to D7). On D8, 50 mg OPC was administered with a single dose of 25 mg warfarin.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form before any study-specific screening procedure was performed,
* Male or female subjects aged 18 to 45 years, inclusive,
* Body mass index (BMI) between 18 and 30 kg/m2,
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead electrocardiogram (ECG),
* Negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies and anti-human immunodeficiency virus (HIV) antibodies at screening,
* Clinical laboratory test results clinically acceptable at screening and at admission to each inpatient period,
* Negative screen for alcohol and drugs of abuse at screening and at admission to each inpatient period,
* Non-smokers or ex-smokers for at least 3 months,
* Able to participate, and willing to give written informed consent and comply with the study restrictions,
* Able to swallow a high number of capsules within a short time frame,

If female:

* Was not of childbearing potential by reason of surgery or, if of childbearing potential, used an effective non-hormonal method of contraception (intrauterine device or intrauterine system; condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he was the sole partner of that subject) for the entire duration of the study,
* Negative serum pregnancy test at screening and a negative urine pregnancy test at admission to each inpatient period.

Exclusion Criteria:

* Any clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders, or had a clinically relevant surgical history,
* Any personal or family history of haemostatic disorder,
* Any personal or family history of bleeding complications after surgery or tooth extraction, nose or gingival bleeding, or haemorrhagic diathesis,
* Any clinically relevant findings in the laboratory tests, particularly any abnormality in the coagulation tests or the liver function tests,
* History of relevant atopy or drug hypersensitivity,
* History of alcoholism and/or drug abuse,
* Current consumption of more than 14 units of alcohol per week [1 unit of alcohol = 280 mL beer (3-4°) = 100 mL wine (10-12°) = 30 mL spirits (40°)],
* Any significant infection or known inflammatory process on screening or admission to each treatment period; any acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period,
* Use of medicines within 2 weeks of admission to first period that could affect the subject's safety or other study assessments, in the investigator's opinion, or intake of any of the prohibited medications (i.e., CYP2C9 inhibitor taken within 1 week prior to start of administration of study drug, and CYP2C9 inducer taken within 4 weeks prior to dosing),
* Previous use of opicapone,
* Use of any investigational drug or participation in any clinical trial within 3 months prior to screening; participation in more than 2 clinical trials within the 12 months prior to screening,
* Blood donation or receipt of any blood transfusion or any blood products within the 3 months prior to screening,
* Vegetarian, vegan or had medical dietary restrictions,
* Not able to communicate reliably with the investigator,
* Unlikely to co-operate with the requirements of the study,
* Unwilling or unable to give written informed consent,
* CYP2C9 poor metaboliser, as assessed by genotyping,

If female:

* Pregnant or breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
R- and S-warfarin plasma concentration | pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post-warfarin

SECONDARY OUTCOMES:
Opicapone plasma concentration | D1 pre-dose, and on D8 at the following time points: pre-dose, 0.5, 2, 4, 6, and 8 h post-opicapone dose
BIA 9-1103 (sulphate metabolite) plasma concentration | D1 pre-dose and from D5 to D7 pre-dose, and on D8 at the following time points: pre-dose, 0.5, 2, 4, 6, 8, 24, 48, 72 and 144 h post-opicapone dose.